

**Study Number: 2022-0776** 

NCT06065449 Page 1 of 12

# Informed Consent/Authorization for Participation in Research

**Title of Research Study:** A Phase III Randomized Trial comparing

Stereotactic Body Radiation Therapy (SBRT) vs Conventional Palliative Radiation Therapy

for Painful Bone Metastases

**Study Number:** 2022-0776

Principal Investigator: Quynh-Nhu Nguyen

Participant's Name Medical Record Number

i artiolpanto i tamo

### **Key Information**

### Why am I being invited to take part in a research study?

You are invited to take part in a research study because you have stable but painful bone metastases (spreading of cancer to the bones) and you may be able to receive palliative radiation therapy as part of your standard treatment. Palliative radiation therapy is radiation therapy intended to treat symptoms (such as pain) instead of the disease itself.

# What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

## Why is this research being done?

The goal of this clinical research study is to compare increasing doses and different treatment schedules of stereotactic body radiation therapy (SBRT) against standard treatment scheduling. SBRT is another type of radiation treatment that gives your doctor the ability to deliver higher doses of radiation to the bone metastases while protecting the normal body tissues.



Researchers want to find the best dose of radiation that is most helpful to patients in relieving symptoms of cancer-related bone pain and improving overall quality of life. Researchers also want to learn if a higher dose of radiation therapy can help decrease the use of drugs to control pain and if it can help to control the disease.

**This is an investigational study.** Radiation therapy in this study is delivered using FDA-approved methods. It is considered investigational to give radiation therapy on different schedules to treat bone metastases.

## How long will the research last and what will I need to do?

You are expected to be in this research study for up to 3 years.

In this study, you will be randomly assigned to a schedule of SBRT (either investigational or standard). After completion of your radiation treatment, you will be asked to follow-up with your treating team after 1 month, then every 3 months for the first year, followed by every 3-6 months after that for up to 3 years total.

Before your study treatment and at each of these study visits, you will be checked for side effects from your radiation treatment, asked about your medication usage to control your pain (if any), have imaging scans, and complete questionnaires asking about the pain, your pain relief, and quality of life.

More detailed information about the study procedures can be found under "What happens if I agree to be in this research?"

# Is there any way being in this study could be bad for me?

Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. If you take part in this study, you may experience side effects affecting your genitals, urinary system, and/or rectum.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

## Will being in this study help me in any way?

Radiation therapy may help to control your pain. Future patients may benefit from what is learned. There may be no benefits for you in this study. It cannot be promised that there will be benefits to you or others.



### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

Instead of being in this research study, you may choose to receive other investigational therapy (if available), palliative radiation as part of your standard of care, or to forego radiation treatment all together in pursuit of alternative treatment for your pain. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer

These alternative treatments have risks and benefits that may be the same or different than those in this research study. The study doctor can discuss these alternative treatments, including their risks and benefits with you.

Your alternative to participating in this research study is to not participate.



## **Detailed Information**

The following is more detailed information about this study in addition to the information listed above.

### Who can I talk to if I have questions or concerns?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team PI, Dr. Quynh-Nhu Nguyen, at 713-563-2300.

This research has been reviewed and approved by an Institutional Review Board (IRB – an ethics committee that reviews research studies). You may talk to them at (713) 792-6477 or IRB Help@mdanderson.org if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

#### How many people will be in this study?

It is expected about 220 people at MD Anderson will be enrolled in this research study.

## What happens if I agree to be in this research?

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will be performed to help the doctor decide if you are eligible:

- You will have a physical exam.
- You will have imaging scans to check the status of the disease. The study doctor
  will decide which type of scan(s) you will have. The types of scans performed
  include: X-rays, a bone scan, computed tomography (CT) scan, positron
  emission tomography/computed tomography (PET/CT) scan, prostate specific
  membrane antigen (PSMA) scan, or magnetic resonance imaging (MRI).
- You will complete questionnaires about your pain, your pain relief, and your quality of life. Completing these questionnaires should take about 15-30 minutes.
- You will be asked about pain medication used (if any) to help control your pain.
- If you can become pregnant, as part of your standard of care, you will have a
  pregnancy test.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.



#### **Study Groups**

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. You will have an equal chance of being assigned to either group.

- If you are in **Group 1**, you will receive either 1 radiation treatment a day for 3 days in a row (not counting weekends or holidays), or you will receive 1 radiation treatment given on 1 day.
- If you are **in Group 2**, you will receive either 1 radiation treatment a day for 5 days, or 1 radiation treatment given on 1 day.

If you are selected for Group 1, the radiation treatment you receive will be determined by the size of the disease being treated. If selected for Group 2, your radiation treatment will be decided based on what your radiation oncologist thinks is in your best interest.

#### **Radiation Therapy**

In order to receive radiation, you will undergo a CT simulation scan. This scan involves lying on a flat table in the exact position you will be in when you receive your treatment. In order to ensure your head and neck do not move, you will wear a custom head and neck mask.

During radiation, you will be asked to lie still for about 30-45 minutes while wearing your mask. You will have a CT scan to make sure you are in the right position before treatment starts. The radiation treatment itself will take about 5-10 minutes to complete each time.

You will no longer be able to receive radiation therapy if intolerable side effects occur or if you are unable to follow study directions.

During the course of your assigned radiation treatment, you will meet with your treating radiation oncologist on a weekly basis to check for any complications or side effects of your treatment.

#### **Follow-Up Visits**

You will be followed up by your research/treatment team by either virtual visit with video or phone calls, or in person clinic visits at the following time points:

- 1 month after your radiation completion (+/- 1 week)
- 3, 6, 9 and 12 months after radiation completion (+/- 4 weeks)
- Every 3-6 months after that for up to 3 years total

At Months 1, 3, 6, 9, 12 and then every 3-6 months after that for up to 3 years:



- Your pain medication usage will be checked/confirmed and you will be asked about your current medication (if any) used to control your pain.
- You will complete questionnaires about your pain, pain relief, and your quality
  of life. The questionnaires can be completed in person during a clinic visit, by
  mail, or by telephone (virtual visits).

At Months 3, 6, 9, 12 and every 3-6 months after the start of radiation therapy, you will have imaging scans (such as X-rays, a bone scan, PET/CT scan, CT scan, PSMA, or MRI) to check the status of the disease per standard of care.

### What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for:

- Completing questionnaires coordinated with your study visits.
- Reporting your side effects experienced to your treating doctor and research team
- Coming to all scheduled visits for follow-up with the research team.

#### What happens if I say yes, but I change my mind later?

You can leave the research at any time; it will not be held against you.

If you withdraw from this study, you can still choose to be treated at MD Anderson. Talk to the study staff first, as it may be dangerous to suddenly stop participation.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

If you decide to withdraw from the trial, you may be asked to explain the extent of your withdrawal. You may choose to forgo follow-up procedures while allowing for your research team to continue data collection from your future standard of care appointments or decide that you would like for no further information to be collected from you all together.

# Is there any way being in this study could be bad for me? (Detailed Risks)

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.



Tell the study staff about any side effects you may have, even if you do not think they are related to the study treatment and procedures.

#### **Radiation Therapy Side Effects**

It is not known how often the side effects of radiation therapy may occur.

| <ul> <li>swelling</li> <li>swelling of the arms or torso</li> <li>skin changes (possible dryness, itching, peeling, and/or blistering</li> <li>hair loss at the treatment site</li> </ul> | <ul> <li>mouth problems</li> <li>trouble swallowing</li> <li>nausea</li> <li>vomiting</li> <li>diarrhea</li> <li>rectal pain and/or bleeding</li> <li>loss of bowel control</li> </ul> | <ul> <li>urinary and/or bladder changes</li> <li>sexual changes</li> <li>inability to produce children</li> <li>joint problems</li> <li>secondary cancers</li> </ul> |
|---|---|---|
|---|---|---|

Radiation therapy may cause you to develop another type of cancer. Side effects may not occur for up to 6 months after radiation therapy is over. Side effects will vary depending on what part of the body is receiving radiation therapy.

#### **Other Risks**

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaires, you are encouraged to contact your doctor or the study chair.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**.

You will be told about any new information that may affect your health, welfare, or choice to stay in the research.

This study may involve unpredictable risks to the participants.

#### **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Getting pregnant will result in your removal from this study.



# Will it cost anything to be in this study? Will I be paid to be in this study?

You and/or your insurance provider will be responsible for the cost of radiation therapy given in this study.

Certain tests and/or procedures that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

You will not receive any compensation for taking part in this study.

#### What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who need to review this information. Complete secrecy cannot be promised. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

Any personal information that could identify you will be removed or changed before data are shared with other researchers or results are made public.

The sponsor, monitors, auditors, the IRB, and the Food and Drug Administration will be granted direct access to your medical records to conduct and oversee the research. By signing this document, you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

Federal law provides additional protections of your medical records and related health information. These are described below.

## Will my data be used for future research?

Your personal information will be collected as part of this study. This data may be used by researchers at MD Anderson, or shared with other researchers and/or institutions for use in future research.

In some cases, all of your identifying information may not be removed before your data are used for future research. If future research is performed at MD Anderson, the



researchers must get approval from the MD Anderson IRB before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

If identifiers are removed from your identifiable private information that is collected during this research, that information could be used for future research studies or shared with another researcher for future research studies without your additional informed consent.

#### Can I be removed from the research study without my permission?

The person in charge of the research study or the sponsor can remove you from the research study without your approval. Possible reasons for removal include intolerance to radiation treatment, severe side effects from your radiation that would stop you from completing your treatment, not following study directions, and not coming to study visits.

#### What happens if I get hurt from being in this study?

If you get sick or hurt and it is related to your participation in this study, you will be given care at MD Anderson (if you are at the clinic when you are sick or hurt). If you get hurt or sick and you are not at the clinic (for example, you are at home or at another doctor's office):

- call your personal doctor right away (or in an emergency, call 911)
- tell your personal doctor or ER staff that you are in this study (try to give them a copy of this consent form or show them your participant card)
- call the study doctor (Dr. Quynh-Nhu Nguyen, at 713-563-2300) or a member of your research team.

You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. Costs of treatment received because you were hurt or sick will be billed to you or your insurance company. No other form of payment is available.

You may also contact the MD Anderson IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

#### What else do I need to know?

MD Anderson may benefit from your participation and/or what is learned in this study.

Your information (both identifiable and de-identified) may be used to create products or to deliver services, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.



# Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.



#### **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| SIGNATURE OF PARTICIPANT | DATE |
|---|---|
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performance. | ormed under this |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAW A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE AIR) |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT | |
| I have discussed this research study with the participant and/or representative, using language that is understandable and appel have fully informed this participant of the nature of this study are and risks and that the participant understood this explanation. | ropriate. I believe that I |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |





## **TRANSLATOR**

| I have translated the above | informed consent as written (without add | litions or |
|---|---|---|
| subtractions) into | and assisted | and assisted the people |
| (Nam | e of Language) | |
| obtaining and providing conscious consent process for this part | sent by translating all questions and resp<br>ticipant. | oonses during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| | translator was a member of the research<br>an the translator, must sign the witness l | ` |